CLINICAL TRIAL: NCT01875666
Title: Defining the HER2 Positive (+) Breast Cancer Kinome Response to Trastuzumab, Pertuzumab, Combination Trastuzumab +Pertuzumab, or Combination Trastuzumab + Lapatinib
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Susan G. Komen Breast Cancer Foundation (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC 1214
Record Dates: First submitted 2013-06-04; First posted 2013-06-12 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-07

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; Kinome; HER two positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Trastuzumab (Active Comparator): single dose intravenous infusion administration of trastuzumab (8 mg/kg)
  Interventions: Drug: Trastuzumab
- pertuzumab (Active Comparator): single dose infusion of pertuzumab (840 mg)
  Interventions: Drug: pertuzumab
- trastuzumab plus pertuzumab (Active Comparator): single dose infusion of combination trastuzumab (8 mg/kg) plus pertuzumab (840 mg)
  Interventions: Drug: Trastuzumab; Drug: pertuzumab
- trastuzumab plus lapatinib (Active Comparator): combination of single dose infusion of trastuzumab (8 mg/kg) plus oral lapatinib (1000 mg daily for 7 days)
  Interventions: Drug: Trastuzumab; Drug: lapatinib

INTERVENTIONS:
Drug: Trastuzumab — 8 mg/kg IV, single dose
  Other Names: Herceptin
  Arms: Trastuzumab; trastuzumab plus lapatinib; trastuzumab plus pertuzumab
Drug: pertuzumab — 840 mg IV single dose
  Other Names: Perjeta
  Arms: pertuzumab; trastuzumab plus pertuzumab
Drug: lapatinib — 1000 mg daily for 7 days
  Other Names: Tykerb
  Arms: trastuzumab plus lapatinib

SUMMARY:
Kinases are a group of proteins that are important in how cancer cells grow. HER2 is a kind of kinase. This study looks at a new approach to identifying kinases, which may help target therapy more precisely.

LCCC1214 is a randomized, multiarm, multicenter, open-label window trial designed to explore the kinome response in Stage I-IV HER2 positive (HER2+) breast cancer patients scheduled to undergo definitive surgery (either lumpectomy, mastectomy or surgical resection of oligometastatic disease). Patients will initiate dosing with either a single HER2-directed agent or a combination of two HER2-directed agents, one week prior to surgery. Forty patients will be randomized to one of four study groups:

A) single dose trastuzumab; B) single dose pertuzumab; C) combination single dose trastuzumab plus single dose pertuzumab; or D) combination single dose trastuzumab plus lapatinib daily for 7 days.

Pre- and post- dosing tissue will be analyzed for kinome response and resistant signatures. The initiation of study drug will be defined by the surgical schedule; there will be no delays in standard treatment for the purposes of this study.

DETAILED DESCRIPTION:
Until recently, our understanding of the kinome has been limited to just 5-10% of the genome-encoded kinases. This limited knowledge prevents a thorough understanding of resistance mechanisms, and precludes individualizing HER2-targeted therapy in HER2+ disease. Fortunately, we have now developed a chemical proteomics approach to define comprehensive kinome activity in cells and tumors (MIB/MS).[1]

We hypothesize that our proteomics approach can be used to characterize the heterogeneity of the kinome activation profiles in HER2+ breast cancer and permit us to identify if adaptive response to HER2 inhibition differs depending on the anti-HER2 drug mechanism of action. This will allow rational prediction of new combinatorial therapies in future clinical trials.

To explore kinome activation in this population, we propose a window trial in stage I-IV HER2+ patients scheduled to undergo definitive surgery (either lumpectomy, mastectomy or surgical resection of oligometastatic disease). Enrolled patients will be randomized to one of four treatment arms; A) single dose trastuzumab; B) single dose pertuzumab; C) combination trastuzumab + pertuzumab for one dose each; or D) combination single dose trastuzumab plus lapatinib daily for one week.

Dosing in each arm will be initiated 7 days prior to surgery, with pre- and post-dosing tissue samples analyzed for kinome response and resistant signatures. To ensure adequate levels of trastuzumab and pertuzumab at the time of surgery, a loading dose of each agent (8 mg/kg IV for trastuzumab, and 840 mg IV fixed dose for pertuzumab) were chosen. The dose of lapatinib was based on prior studies of lapatinib administered in combination with trastuzumab. Given the varied pharmacokinetic profiles of the three agents and limited dosing, we expect exposure levels of the agents to be different relative to respective steady state levels. Therefore qualitative rather than quantitative measures will be key.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent
* Age >/= 18 years
* Histologically confirmed HER2+ breast cancer: IHC 3+ or fluorescence in situ hybridization [FISH] amplified; by clinical assay on either primary or metastatic tumor
* Stage I-IV disease

  * For patients with Stage I-IIIc disease:

    1. Scheduled for lumpectomy or mastectomy
    2. No prior or current therapy for breast cancer
    3. Not considered a candidate for therapeutic neoadjuvant treatment
  * For patients with Stage IV disease:

    1. Scheduled for surgical resection of oligometastatic disease
    2. Previously untreated for breast cancer
* Normal relevant end organ function as defined by the following:

  * ANC>1500 cells/mL
  * Platelets > 100,000 cells/mL
  * Hemoglobin > 10 g/dL
  * Total bilirubin ≤ 1.5 x ULN (unless known Gilbert's syndrome)
  * AST and ALT ≤ 2.5 X ULN
  * Creatinine ≤ 1.5 X ULN OR Calculated creatinine clearance ≥50 mL/min OR 24-hour urine creatinine clearance ≥50 mL/min
  * Left Ventricular Ejection Fraction ≥ 50% by ECHO (preferred) or MUGA
* For women of childbearing potential, agreement to use an effective form of contraception (patient and/or partner, e.g., surgical sterilization, a reliable barrier method, birth control pills, or contraceptive hormone implants) and to continue its use for the duration of the study treatment, and for a minimum of 6 months following trastuzumab and/or pertuzumab administration.
* Sufficient fresh or frozen tissue remaining from pre-treatment core biopsy/ incisional biopsy or willing to undergo biopsy (at UNC via LCCC9819) for research purposes only (approximately 10mg or one core's worth of tissue needed)
* Surgeon and medical oncologist agree one week window trial is appropriate/safe for the patient and that surgery appointment can accommodate treatment schedule as outlined in the study schema (section 4.1).
* UNC patients must co-enroll into LCCC9819 for collection of tissue samples

Exclusion Criteria:

* Pregnant or lactating female
* Prior radiation therapy to the target lesion
* Use of any investigational drug within 28 days or five half-lives, whichever is shorter, prior to the first dose of study medication; a minimum of 10 days between termination of the investigational drug and treatment with study medication is required
* Any major radiotherapy, tumor-directed systemic or immunotherapy within the last 4 weeks for any indication
* Candidate for therapeutic neoadjuvant treatment
* Active infection
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease)
* Required administration of concomitant moderate or strong inhibitors or inducers of CYP3A4 for 14 days prior to the first dose of study drug prior amiodarone for up to 6 months prior to day 1 of study treatment
* Inability to take oral medications e.g., impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral medications (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* History or evidence of cardiovascular risk including any of the following:

  * Current uncontrolled hypertension (systolic >150 mm Hg and/or diastolic >100 mmHg) or unstable angina
  * History of serious cardiac arrhythmia requiring treatment (exceptions: atrial fibrillation, paroxysmal supraventricular tachycardia)
  * History of myocardial infarction within 6 months of day 1 of dosing
  * History of CHF of New York Heart Association (NYHA) criteria
* Known human immunodeficiency virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection which will be allowed)
* Have acute or currently active/requiring anti-viral therapy hepatic or biliary disease (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol
* Any other concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
difference in kinome activation pre and post treatment | 7-10 days prior to surgery and at surgery
  To identify differential kinome activation before and after treatment with a single dose of trastuzumab, pertuzumab, the combination of trastuzumab + pertuzumab, or the combination of single dose trastuzumab+once daily lapatinib for 7 days, in patients with HER2+ breast cancer

SECONDARY OUTCOMES:
predictability in kinome activation | kinoming analysis of tissue will be done after subject participation, which will last from 7-10 days prior to surgery.
  to see if different kinase activation patterns can predict the optimal HER2 inhibition for treatment.

OTHER OUTCOMES:
number and type of adverse reactions | subjects will be followed for AEs during the one week to 10 days (mode expected to be 7 days) prior to surgery
  Documentation of adverse events according to CTCAE criteria.
future predictive molecular markers in response to each treatment | one year
  Identification of molecular markers correlated with drug administration for each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Carey, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - IU Simon Cancer Center, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - MD Anderson, Houston, Texas